CLINICAL TRIAL: NCT03216109
Title: Improving Supportive Care For Patients With Thoracic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Carevive Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Manali Patel, Principal Investigator Staff Oncologist VAPAHCS, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PAT0001ARG
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; Quality of Life; Supportive Care
Keywords: Supportive Care; Quality of Life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly telephone symptom assessment (Experimental): Each patient who is enrolled in the intervention will receive a weekly phone call from the Research Assistant for a total of 9 months to assess symptoms using the Edmonton Symptom Assessment Scale. Results of the symptom assessments will be provided to the clinic staff (RN and MD) for review each week. Symptom assessments will be documented into an encrypted, HIPAA compliant digital platform which provides longitudinal symptom data management and also provides symptom assessment tools for the clinical team in their intervention strategies.
  In addition, patients will complete symptom and quality of life surveys at 0, 3, 6 and 9 months.
  Interventions: Behavioral: Weekly telephone symptom assessment
- Control Arm (No Intervention): Patients randomized to usual clinical care will receive standard of care for thoracic malignancies as provided by the VA Palo Alto Health Care System. Patients will complete outcome surveys at 0, 3, 6, and 9 months.

INTERVENTIONS:
Behavioral: Weekly telephone symptom assessment — Each patient who is enrolled in the intervention will receive a weekly phone call from the Research Assistant for a total of 9 months to assess symptoms using the Edmonton Symptom Assessment Scale. Results of the symptom assessments will be provided to the clinic staff (RN and MD) for review each week. Care plans will be generated using an electronic management platform
  Arms: Weekly telephone symptom assessment

SUMMARY:
The purpose of this study is to use a proactive approach to improve symptom management of patients with thoracic malignancies and ensure receipt of evidence-based cancer care delivery. In this pilot study, the investigators propose to evaluate the feasibility of using outbound, proactive telephone symptom assessment strategies and ensuring evidence-based care receipt and measure the efficacy of this approach on patient satisfaction with their care, patient activation, quality of life and use of healthcare resources.

DETAILED DESCRIPTION:
The investigators have previously shown in previous work that patients and caregivers who experience thoracic malignancies express poor symptom management that result in utilization of healthcare resources after-hours for symptoms that could have been prevented if assessed more proactively and prospectively. Currently, there are limited proactive approaches to prospectively identify and intervene on patient-reported symptoms. The purpose of this study is to enhance symptom assessment strategies by using a proactive assessment approach to improve symptom relief for patients with thoracic malignancies.

The investigators will test whether a proactive telephone symptom assessment and management strategy is feasible and can facilitate early patient report of their symptoms and intervention. The knowledge gained from this approach will be used to identify solutions that can be scaled nationally to improve patient-reported symptom management and patient satisfaction with their clinical care.

ELIGIBILITY:
Inclusion Criteria:

* All patients with lung cancer treated at VA Palo Alto. This includes all newly diagnosed patients and those under follow-up care.

Exclusion Criteria:

* Patients who do not anticipate receiving oncology care at the VA Palo Alto Health Care System.
* Patients who are unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Symptom documentation | 6 months after patient enrollment
  Defined as 75% documentation of symptoms for patients in the intervention arm

SECONDARY OUTCOMES:
Emergency Department Visit (Chart Review) | 9 months after patient enrollment
  Emergency Department visits for each patient will be abstracted by electronic medical record for each patient at 9 months
Hospitalizations (Chart Review) | 9 months after patient enrollment
  Hospitalizations for each patient will be abstracted by electronic medical record for each patient at 9 months
Change in Quality of Life using the Functional Assessment of Cancer Therapy - Lung survey | Change in Quality of Life from baseline to month 3
  Each patient will receive a validated survey to assess quality of life at baseline and 3 months
Change in Quality of Life using the Functional Assessment of Cancer Therapy - Lung survey | Change in Quality of Life from baseline to month 6
  Each patient will receive a validated survey to assess quality of life at baseline and 6 months
Change in Quality of Life using the Functional Assessment of Cancer Therapy - Lung survey | Change in Quality of Life from baseline to month 9
  Each patient will receive a validated survey to assess quality of life at baseline and 9 months
Change in patient satisfaction with decision-making using the Satisfaction with Decision Survey | Change in patient satisfaction with decision--making from baseline to 3 months
  Each patient will receive a validated survey to assess their satisfaction with decision at baseline and 3 months
Change in patient satisfaction with decision-making using the Satisfaction with Decision Survey | Change in patient satisfaction with decision--making from baseline to 6 months
  Each patient will receive a validated survey to assess their satisfaction with decision at baseline and 6 months
Change in patient satisfaction with decision-making using the Satisfaction with Decision Survey | Change in patient satisfaction with decision--making from baseline to 9 months
  Each patient will receive a validated survey to assess their satisfaction with decision at baseline and 9 months
Change in Patient Activation using the validated Patient Activation Measure | Change in patient activation from baseline to 3 months
  Each patient will receive a validated survey to assess their activation at baseline and 3 months
Change in Patient Activation using the validated Patient Activation Measure | Change in patient activation from baseline to 6 months
  Each patient will receive a validated survey to assess their activation at baseline and 6 months
Change in Patient Activation using the validated Patient Activation Measure | Change in patient activation from baseline to 9 months
  Each patient will receive a validated survey to assess their activation at baseline and 9 months
Change in symptoms using the validated Edmonton Symptom Assessment Scale | Change in symptoms from baseline to 3 months
  Each patient will receive a validated survey to assess their symptoms at baseline and 3 months
Change in symptoms using the validated Edmonton Symptom Assessment Scale | Change in symptoms from baseline to 6 months
  Each patient will receive a validated survey to assess their symptoms at baseline and 6 months
Change in symptoms using the validated Edmonton Symptom Assessment Scale | Change in symptoms from baseline to 9 months
  Each patient will receive a validated survey to assess their symptoms at baseline and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Manali I Patel, MD, Principal Investigator — Faculty
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banks LC, Kapphahn K, Das M, Patel MI. Randomized Trial of a Volunteer-Led Symptom Assessment Intervention on Documentation, Patient-Reported Outcomes, and Health Care Use Among Veterans With Lung Cancer. JCO Oncol Pract. 2024 Mar;20(3):419-428. doi: 10.1200/OP.23.00557. Epub 2024 Jan 11. PMID 38207246
- [Derived] Patel MI, Banks L, Das M. Improving supportive care for patients with Thoracic Malignancies - A randomized controlled trial. Contemp Clin Trials Commun. 2022 May 27;28:100929. doi: 10.1016/j.conctc.2022.100929. eCollection 2022 Aug. PMID 35669484